CLINICAL TRIAL: NCT00786292
Title: Evaluation of Variable Pressure Support Ventilation in the Therapy of Acute Lung Injury (EVA-Trial)
Brief Title: Evaluation of Variable Pressure Support Ventilation in the Therapy of Acute Lung Injury
Acronym: EVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, PD Dr. Marcelo Gama de Abreu, Prof. Dr., Technische Universität Dresden
Purpose: Treatment
Other Study IDs: EK276112007
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2009-07

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noisy PSV (Other): Assisted mechanical ventilation with noisy PSV
  Interventions: Other: Assisted mechanical ventilation
- PSV (Other): Assisted mechanical ventilation with PSV
  Interventions: Other: Assisted mechanical ventilation

INTERVENTIONS:
Other: Assisted mechanical ventilation — Patients will be mechanically ventilated with noisy PSV and PSV in random sequence

SUMMARY:
Variable pressure support during assisted spontaneous breathing (noisy PSV) has been shown to improve the respiratory function in experimental acute lung injury (ALI). We aimed at comparing the effects of noisy PSV with traditional PSV on the respiratory function of patients suffering from ALI.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 75 yrs
* 150 mmHg < PaO2/FIO2 < 300 mmHg
* mechanical ventilation with PSV or BIPAP
* less than 15 days of mechanical ventilation
* at least 20% of minute ventilation originated from spontaneous breathing

Exclusion Criteria:

* BMI > 35
* esophageal disease
* neuromuscular disease
* instable thorax
* pneumothorax
* head trauma
* brain injury
* increased intracranial pressure
* agitation
* increased need for vasoactive drugs
* chronic lung disease
* acute coronary disease
* participation in another clinical trial within the last 4 weeks at enrollment

Interruption criteria:

* acute change of mental status
* SaO2 < 92%
* pHa < 7.30
* respiratory rate > 30 or < 6 /min
* dyspnea
* diaphragm/thorax antagonism
* diaphoresis
* abnormal use of respiratory muscles
* increase of the heart rate above 120% of baseline or absolute value < 60 or > 130 /min
* mean arterial pressure above 120% of baseline or absolute value < 70 or > 110 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Effect on the arterial oxygenation

SECONDARY OUTCOMES:
Effect on the work of breathing
Effect on PaCO2

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Gama de Abreu, MD, PhD, Principal Investigator — Department of Anesthesiology, University Clinic Carl Gustav Carus, Technical University Dresden
Locations (1):
- University Clinic Carl Gustav Carus, Technical University Dresden, Dresden, Germany

REFERENCES:
- [Derived] Spieth PM, Guldner A, Huhle R, Beda A, Bluth T, Schreiter D, Ragaller M, Gottschlich B, Kiss T, Jaber S, Pelosi P, Koch T, Gama de Abreu M. Short-term effects of noisy pressure support ventilation in patients with acute hypoxemic respiratory failure. Crit Care. 2013 Oct 31;17(5):R261. doi: 10.1186/cc13091. PMID 24172538